CLINICAL TRIAL: NCT06998524
Title: A Phase III, Multicenter, Open-Label Study to Evaluate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Emicizumab Prophylaxis in Patients With Type 3 Von Willebrand Disease
Brief Title: A Study to Assess the Efficacy and Safety of Emicizumab in Participants With Type 3 Von Willebrand Disease
Acronym: WILL-EMI
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WP45338; 2024-515622-80-00 (EU CTIS Number)
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Von Willebrand Disease, Type 3
MeSH Terms: conditions — von Willebrand Disease, Type 3 | interventions — emicizumab; von Willebrand Factor; Factor VIII

STUDY DESIGN:
Intervention Model Description: Participants on prior SOC on-demand therapy will be randomized into Arms A and B. Participants on prior SOC prophylactic therapy, who participated in the NIS WP45335 (NCT06883240) and meet the eligibility criteria for this study, will be enrolled into Arm C.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A (Prior On-Demand SOC): Emicizumab Prophylaxis for 24 Weeks (Experimental): Participants who are randomized to Arm A, taking on-demand standard of care (SOC) treatment at the time of study entry (and for at least 24 weeks prior to enrollment), will receive emicizumab SC prophylaxis.
  Interventions: Drug: Emicizumab
- Arm B (Prior On-Demand SOC): On-Demand SOC for 24 Weeks (Active Comparator): Participants who are randomized to Arm B, taking on-demand standard of care (SOC) treatment at the time of study entry (and for at least 24 weeks prior to enrollment), will continue to receive their current SOC on-demand treatment until Week 24.
  Interventions: Drug: von Willebrand Factor (VWF) Concentrates; Drug: Factor VIII (FVIII) Concentrates; Drug: von Willebrand Factor (VWF) and Factor VIII (FVIII) Concentrates; Drug: Bypassing Agents
- Arm C (Prior Prophylaxis SOC): Emicizumab Prophylaxis for 24 Weeks (Experimental): Participants who enroll in Arm C, taking SOC prophylactic treatment at the time of study entry and for at least 24 weeks of observation during the preceding NIS WP45335, will receive emicizumab SC prophylaxis.
  Interventions: Drug: Emicizumab
- Treatment Extension Period for All Arms: Emicizumab Prophylaxis (Experimental): Participants in Arms A and C who have completed 24 weeks of emicizumab prophylaxis and who derive benefit from emicizumab will have the opportunity to continue to receive emicizumab prophylaxis in the extension period. Participants in Arm B who have completed 24 weeks of SOC on-demand treatment will have the opportunity to receive emicizumab prophylaxis in the extension period.
  Interventions: Drug: Emicizumab

INTERVENTIONS:
Drug: Emicizumab — Participants will receive emicizumab 3 milligrams per kilogram (mg/kg) subcutaneous (SC) injections every week (QW) for the first 4 weeks as loading doses, followed by maintenance doses of emicizumab 3 mg/kg SC once every 2 weeks (Q2W).
  During the extension period, participants may remain on maintenance dose of emicizumab 3 mg/kg Q2W, or change their emicizumab maintenance regimen to 1.5 mg/kg once every week (QW) or 6 mg/kg once every 4 weeks (Q4W), if they prefer and if agreed by the investigators.
  Other Names: Hemlibra; RO5534262; RG6013
  Arms: Arm A (Prior On-Demand SOC): Emicizumab Prophylaxis for 24 Weeks; Arm C (Prior Prophylaxis SOC): Emicizumab Prophylaxis for 24 Weeks; Treatment Extension Period for All Arms: Emicizumab Prophylaxis
Drug: von Willebrand Factor (VWF) Concentrates — Used according to local labeling or local treatment guidelines.
  Arms: Arm B (Prior On-Demand SOC): On-Demand SOC for 24 Weeks
Drug: Factor VIII (FVIII) Concentrates — Used according to local labeling or local treatment guidelines.
  Arms: Arm B (Prior On-Demand SOC): On-Demand SOC for 24 Weeks
Drug: von Willebrand Factor (VWF) and Factor VIII (FVIII) Concentrates — Used according to local labeling or local treatment guidelines.
  Arms: Arm B (Prior On-Demand SOC): On-Demand SOC for 24 Weeks
Drug: Bypassing Agents — Used according to local labeling or local treatment guidelines.
  Arms: Arm B (Prior On-Demand SOC): On-Demand SOC for 24 Weeks

SUMMARY:
This is a Phase III, multicenter, open-label clinical study designed to evaluate the efficacy, safety, pharmacokinetics, and pharmacodynamics of emicizumab prophylaxis in participants aged 1 month and above, who have been diagnosed with Type 3 von Willebrand disease (VWD). Participants on prior standard of care (SOC) on-demand therapy will be assessed via a randomized comparison (Arm A - emicizumab prophylaxis and Arm B - continuation of SOC on-demand therapy), while participants on prior SOC prophylactic therapy (Arm C - emicizumab prophylaxis) will be assessed via intra-participant analysis with data obtained from the preceding non-interventional study (NIS), WP45335 (NCT06883240).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Type 3 von Willebrand disease (VWD), based on medical records
* Preexisting medical record verifying the status of von Willebrand factor (VWF) inhibitor (positive or negative, including titer if available)
* Adequate hematologic, hepatic, and renal function
* For participants of childbearing potential: agreement to remain abstinent or adhere to the contraception requirements

Additional Inclusion Criteria for Arms A and B:

* Age ≥1 month at the time of signing Informed Consent/Assent Form
* Documented previous use of on-demand therapy with intermittent (less than once a week) on-demand SOC therapy for VWD
* Having ≥2 treated bleeds (except menstrual bleeds) with factor concentrate within 24 weeks prior to enrollment

Additional Inclusion Criteria for Arm C:

* Age ≥2 years at the time of signing Informed Consent/Assent Form
* Documented and confirmed previous use of SOC prophylactic therapy for VWD (1-3 times weekly, as per prescribed dose) as described in the eligibility of Study WP45335
* Have completed all study requirements as defined in the WP45335 protocol for at least 24 weeks

Exclusion Criteria:

* Inherited or acquired bleeding disorder other than Congenital Type 3 VWD
* History of gastrointestinal bleeding within 18 months prior to enrollment, or any previous diagnosis of angiodysplasia
* History of intracranial hemorrhage
* Previous or current treatment for thromboembolic disease or signs of thromboembolic disease
* Other conditions (e.g., certain autoimmune diseases) that may increase risk of bleeding or thrombosis
* History of clinically significant hypersensitivity associated with monoclonal antibody therapies or components of the emicizumab injection
* Use of systemic immunomodulators (e.g., interferon) at enrollment or planned use during the study, with the exception of anti-retroviral therapy

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Annualized Bleed Rate (ABR) for Treated Bleeds in the Randomized Arms | From Baseline to at least 24 weeks

SECONDARY OUTCOMES:
ABR for All Bleeds in the Randomized Arms | From Baseline to at least 24 weeks
ABR for Treated Spontaneous Bleeds in the Randomized Arms | From Baseline to at least 24 weeks
ABR for Treated Joint Bleeds in the Randomized Arms | From Baseline to at least 24 weeks
Intra-Participant Comparison of the ABR for Treated Bleeds with Prophylactic Emicizumab Versus Prophylactic SOC from the Preceeding Non-Interventional Study (NIS) WP45335 | From Baseline to at least 24 weeks
Intra-Participant Comparison of the ABR for All Bleeds with Prophylactic Emicizumab Versus Prophylactic SOC from the Preceeding NIS WP45335 | From Baseline to at least 24 weeks
Intra-Participant Comparison of the ABR for Treated Spontaneous Bleeds with Prophylactic Emicizumab Versus Prophylactic SOC from the Preceeding NIS WP45335 | From Baseline to at least 24 weeks
Intra-Participant Comparison of the ABR for Treated Joint Bleeds with Prophylactic Emicizumab Versus Prophylactic SOC from the Preceeding NIS WP45335 | From Baseline to at least 24 weeks
Incidence and Severity of Adverse Events, with Severity Determined According to the World Health Organization (WHO) Toxicity Grading Scale | From first dose of study treatment until 24 weeks after final dose of study treatment (up to 3 years, 11 months)
Incidence and Severity of Thromboembolic Events | From first dose of study treatment until 24 weeks after final dose of study treatment (up to 3 years, 11 months)
Incidence and Severity of Thrombotic Microangiopathy Events | From first dose of study treatment until 24 weeks after final dose of study treatment (up to 3 years, 11 months)
Incidence and Severity of Injection-Site Reactions | From first dose of study treatment until 24 weeks after final dose of study treatment (up to 3 years, 11 months)
Incidence of Adverse Events Leading to Drug Discontinuation | From first dose of study treatment until 24 weeks after final dose of study treatment (up to 3 years, 11 months)
Incidence of Severe Hypersensitivity, Anaphylaxis, or Anaphylactoid Reactions | From first dose of study treatment until 24 weeks after final dose of study treatment (up to 3 years, 11 months)
Incidence of Clinical Laboratory Abnormalities | From first dose of study treatment until 24 weeks after final dose of study treatment (up to 3 years, 11 months)
Trough Plasma Concentration of Emicizumab at Prespecified Timepoints During the Treatment Period | Predose and at prespecified timepoints from first dose of emicizumab until study completion (up to 3 years, 11 months)
Percentage of Participants with Anti-Drug Antibodies (ADAs) to Emicizumab at Baseline and with ADAs to Emicizumab During the Treatment Period | Baseline and at prespecified timepoints from first dose of emicizumab until study completion (up to 3 years, 11 months)
Change from Baseline in Respiratory Rate Over Time | Baseline, Weeks 1, 2, 25, and every 12 weeks thereafter (weeks after switch to emicizumab for Arm B only) until study completion (up to 3 years, 11 months)
Change from Baseline in Pulse Rate Over Time | Baseline, Weeks 1, 2, 25, and every 12 weeks thereafter (weeks after switch to emicizumab for Arm B only) until study completion (up to 3 years, 11 months)
Change from Baseline in Systolic Blood Pressure Over Time | Baseline, Weeks 1, 2, 25, and every 12 weeks thereafter (weeks after switch to emicizumab for Arm B only) until study completion (up to 3 years, 11 months)
Change from Baseline in Diastolic Blood Pressure Over Time | Baseline, Weeks 1, 2, 25, and every 12 weeks thereafter (weeks after switch to emicizumab for Arm B only) until study completion (up to 3 years, 11 months)
Change from Baseline in Body Temperature Over Time | Baseline, Weeks 1, 2, 25, and every 12 weeks thereafter (weeks after switch to emicizumab for Arm B only) until study completion (up to 3 years, 11 months)
Change from Baseline in Electrocardiogram (ECG) Parameters Over Time: QT, QTcF, RR, PR, and QRS Intervals | Baseline and study completion (up to 3 years, 11 months)
Change from Baseline in Heart Rate Over Time, as Measured by Electrocardiogram (ECG) | Baseline and study completion (up to 3 years, 11 months)
Change from Baseline in the PROMIS-29 Questionnaire Pain Interference Domain Score Over Time | Baseline and at prespecified timepoints until study completion (up to 3 years, 11 months)
  PROMIS-29 stands for Patient-Reported Outcomes Measurement Information System-29
Change from Baseline in the PROMIS-29 Questionnaire Fatigue Domain Score Over Time | Baseline and at prespecified timepoints until study completion (up to 3 years, 11 months)
  PROMIS-29 stands for Patient-Reported Outcomes Measurement Information System-29

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (26):
- United States (3):
  - UC Davis, Sacramento, California
  - University of Florida, Gainesville, Florida
  - Washington University School of Medicine, St Louis, Missouri
- UZ Leuven Gasthuisberg, Leuven, Belgium
- Canada (2):
  - The Hospital for Sick Children, Toronto, Ontario
  - McGill University Health Center, Montreal, Quebec
- IPS SURA Industriales Medellín, Medellín, Colombia
- France (2):
  - Hopital Claude Huriez - CHU Lille, Lille
  - Groupe Hospitalier Necker Enfants Malades, Paris
- Germany (3):
  - Universitätsklinikum Bonn, Bonn
  - Gerinnungszentrum Rhein-Ruhr;Gerinnungsambulanz, Duisburg
  - Hämophiliezentrum Med. Klinik III/Institut für Transfusionsmedizin, Frankfurt/M.
- Italy (3):
  - Universita' Degli Studi La Sapienza-Ist.Di Ematologia, Rome, Lazio
  - IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - AOU Careggi, Florence, Tuscany
- Japan (2):
  - Kurume University Hospital, Fukuoka
  - Nagoya University Hospital, Nagoya
- Erasmus MC, Rotterdam, Netherlands
- Instytut Hematologii i Transfuzjologii, Warsaw, Poland
- Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg, South Africa
- Spain (2):
  - Hospital Universitario la Paz, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
- Sahlgrenska Universitetssjukhuset, Gothenburg, Sweden
- United Kingdom (3):
  - St Thomas' Hospital, London
  - Great Ormond Street Hospital, London
  - Manchester Royal Infirmary, Manchester

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing